CLINICAL TRIAL: NCT02019004
Title: Treatment of Forehead/Glabellar Rhytide Complex With Onabotulinum Toxin A Versus Incobotulinum Toxin A Injection: A Split-face, Double-blinded, Randomized Control Trial
Brief Title: A Pilot Study Testing Onabotulinum Toxin A Versus Incobotulinum Toxin A Injections for Facial Wrinkles
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU83962
Record Dates: First submitted 2013-11-12; First posted 2013-12-24 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Wrinkles
MeSH Terms: interventions — onabotulinum toxin A; Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Onabotulinum Toxin A (Active Comparator): One side of the face will be randomized to receive Onabotulinum Toxin A injections in the forehead and glabellar region of the face.
  Interventions: Drug: Onabotulinum Toxin A
- Incobotulinum Toxin A (Active Comparator): The other side of the face will be randomized to receive Incobotulinum Toxin A injections in the glabellar and forehead region of the face.
  Interventions: Drug: Incobotulinum Toxin A

INTERVENTIONS:
Drug: Onabotulinum Toxin A
  Other Names: Botox
  Arms: Onabotulinum Toxin A
Drug: Incobotulinum Toxin A
  Other Names: Xeomin
  Arms: Incobotulinum Toxin A

SUMMARY:
The purpose of this study is to compare the effectiveness of Botox® (Onabotulinum Toxin A) versus Xeomin® (incobotulinum toxin A) for the treatment of forehead and glabellar (vertical lines between the eyebrows) wrinkles.

DETAILED DESCRIPTION:
Subjects will be screened, photographed, assessed, and randomized to be injected with onabotulinum toxin A on one side and incobotulinum toxin A on the other side during their first clinic visit. Subjects will return for a 2 week, 2 month, 3 month, 4 month, 5 month, and 6 month follow-up to have photographs taken by the unblinded research assistant at relaxed and full contraction.

This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males
2. In good health
3. Is 20-65 years of age
4. Has static and moderate dynamic forehead/glabellar wrinkles
5. Has willingness and the ability to understand and provide informed consent and communicate with the study staff

Exclusion Criteria:

1. Pregnant or lactating
2. Younger than 20 or older than 65 years of age
3. Has received the following treatments in the forehead or glabellar region:

   1. botulinum toxin injections in the past 6 months
   2. ablative laser procedure in the past 6 months
   3. radiofrequency device treatment in the past 6 months
   4. ultrasound device treatment in the past 6 months
   5. medium to deep chemical peel in the past 6 months
   6. temporary soft tissue augmentation material in the area to be treated in the past year
   7. semi-permanent soft tissue augmentation material in the area to be treated in the past 2 years
   8. permanent soft tissue augmentation material in the area to be treated
4. Is planning to receive within the next 6 months, any cosmetic procedure (such as any chemical peels, botulinum toxin injections, ablative or non-ablative laser procedures, filler injections, radiofrequency procedures, dermabrasion, ultrasound and face lifting procedures) in the forehead or glabellar region.
5. Is planning to use tretinoin or retinoic acid in the next 6 months
6. Has an active infection in the forehead or glabellar region (excluding mild acne)
7. Is allergic to cow's milk protein
8. Is allergic to albumin
9. Taking aminoglycoside
10. Is currently using anticoagulation therapy
11. Has a history of bleeding disorders
12. Has a mental illness
13. Unable to understand the protocol or to give informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in glabellar wrinkle score from baseline to 6 months for botox vs. xeomin | At baseline and at 6 months
  Two blinded dermatologists will rate each photograph of each subject at baseline and at month 6. The glabellar wrinkle rating is:
  0: no facial wrinkles
  1. mild facial wrinkles
  2. moderate facial wrinkles
  3. severe facial wrinkling
Change in forehead wrinkle score from baseline to 6 months for botox vs. xeomin | At baseline and at 6 months
  Two blinded dermatologists will rate each photograph of each subject at baseline and at month 6. The forehead wrinkle Merz rating is:
  0: no wrinkles
  1. minimal wrinkles
  2. mild wrinkles
  3. moderate wrinkles
  4. severe wrinkles

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States